CLINICAL TRIAL: NCT05107856
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation Study of PRT1419 Injection as Monotherapy or in Combination With Azacitidine or Venetoclax in Patients With Relapsed/Refractory Myeloid or B-cell Malignancies
Brief Title: PRT1419 as Monotherapy or in Combination With Azacitidine or Venetoclax in R/R Myeloid or B-cell Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Prelude Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT1419-03
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukemia; B-cell Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Chronic Myelomonocytic Leukemia; Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Small Lymphocytic Lymphoma
Keywords: Acute Myeloid Leukemia (AML); Azacitidine; B-cell Malignancies; B-cell Non-Hodgkin lymphoma; Chronic lymphocytic leukemia (CLL); Chronic Myelomonocytic Leukemia (CMML); Follicular Lymphoma; Hematologic Malignancies; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Myelodysplastic Syndromes (MDS); Myeloid cell leukemia-1 (MCL-1); Myeloproliferative Neoplasm (MPN); PRT1419; Relapsed/Refractory Myeloid; Small lymphocytic lymphoma (SLL); Venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Myelodysplastic Syndromes; Myeloproliferative Disorders; Hematologic Neoplasms; Recurrence | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PRT1419 Monotherapy (Experimental): PRT1419 will be administered by intravenous infusion once weekly on a 28-day treatment cycle at the dose level assigned.
  Interventions: Drug: PRT1419
- PRT1419/Azacitidine Combination (Experimental): PRT1419 will be administered by intravenous infusion once weekly on a 28-day treatment cycle at the dose level assigned and Azacitidine will be administered by intravenous or subcutaneous on Days 1 through 7 (or alternatively on Days 1 through 5, 8 and 9) of each 28-day treatment cycle.
  Interventions: Drug: PRT1419; Drug: Azacitidine
- PRT1419/Venetoclax Combination (Experimental): PRT1419 will be administered by intravenous infusion once weekly on a 28-day treatment cycle at the dose level assigned and Venetoclax will be administered orally after either a 3-day or 5-week ramp-up period to reach 400 mg daily administration, prior to commencing PRT1419 administration.
  Interventions: Drug: PRT1419; Drug: Venetoclax

INTERVENTIONS:
Drug: PRT1419 — PRT1419 will be administered by intravenous infusion
Drug: Azacitidine — Azacitidine will be administered by intravenous or subcutaneous
  Arms: PRT1419/Azacitidine Combination
Drug: Venetoclax — Venetoclax will be administered orally
  Arms: PRT1419/Venetoclax Combination

SUMMARY:
This is a Phase 1 dose-escalation study of PRT1419, a myeloid cell leukemia-1 (MCL-1) inhibitor, in participants with selected relapsed/refractory myeloid or B-cell malignancies. The purpose of this study is to evaluate the safety and tolerability of PRT1419 monotherapy and in combination with either azacitidine or venetoclax, describe any dose limiting toxicities (DLTs), define the dosing schedule, and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation, Phase 1 study of PRT1419, a MCL-1 inhibitor, evaluating participants with acute myeloid leukemia (AML), chronic myelomonocytic leukemia (CMML), myelodysplastic syndrome (MDS), MDS/myeloproliferative neoplasm (MPN) overlap syndrome, chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL), and B-cell non-hodgkin lymphoma (NHL) including marginal zone lymphoma, follicular lymphoma or mantle cell lymphoma. Participants in study will receive PRT1419 as monotherapy or in combination with either Azacitidine (AZA) or Venetoclax (VEN). The study includes multiple dose escalations and expansion cohorts for RP2D confirmation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations (including contraception requirements), and other study procedures
* Refractory/relapsed disease, having progressed on prior treatment, and without access to further approved therapies or ineligible for approved therapies, in one of the following disease categories: AML, CMML, MDS, MDS/MPN Overlap Syndrome, CLL/SLL, and B-cell NHLs
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 to 2
* Adequate organ function (hematology, hepatic, renal, and coagulation)

Exclusion Criteria:

* Active inflammatory disorders of the gastrointestinal tract, a history of bariatric surgery or other disorders with the potential for GI malabsorption
* Cardiac function compromise, as assessed by echocardiogram or protocol-specified biochemical markers of cardiac damage, or protocol-defined clinically significant heart disease
* History of cerebrovascular accident or transient ischemic attack, within 6 months of screening. Participants with a history of pulmonary embolism must not be symptomatic at enrollment
* Undergone hematopoietic stem-cell transplantation (HSCT) within the last 90 days or have graft-versus-host disease (GVHD) Grade > 1 at study entry
* Uncontrolled intercurrent illnesses, poorly controlled hypertension or dyslipidemias, Unstable central nervous system (CNS) metastases
* Treatment with either OATP1B1, OATP1B3 substrates or strong inhibitors of CYP2C8, CYP3A4, and any medication contraindicated in combination with AZA or VEN
* Prior exposure to an MCL-1 inhibitor
* Within 5 half-lives or 14 days (whichever is longer) following the last systemic anti-cancer therapy
* History of another malignancy except for:

  1. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  2. Adequately treated cervical or breast carcinoma in situ without evidence of disease
  3. Asymptomatic prostate cancer without known metastatic disease and no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for >1 year prior to enrollment
  4. Other malignancy treated with curative intent with no known active disease for > 2 years prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) of PRT1419 | Baseline through Day 28
  Dose limiting toxicities will be evaluated over the 28-day observation period
Safety and tolerability of PRT1419: AEs, SAEs, CTCAE assessments | Baseline through approximately 3 years
  Safety and tolerability will be assessed by recording adverse events (AEs), serious adverse events (SAEs), and DLTs according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Maximum tolerated dose (MTD)/Recommended phase 2 dose (RP2D) and schedule of PRT1419 | Baseline through approximately 2 years
  The MTD/RP2D will be established for further investigation in participants with advanced hematologic malignancies

SECONDARY OUTCOMES:
Pharmacokinetic profile of PRT1419 monotherapy and in combination with AZA or VEN: maximum observed plasma concentration | Baseline through approximately 3.5 years
  PRT1419 pharmacokinetics will be calculated by maximum observed plasma concentration
Pharmacokinetic profile of PRT1419 monotherapy and in combination with AZA or VEN: Time to maximal plasma concentration | Baseline through approximately 3.5 years
  PRT1419 pharmacokinetics will be calculated by time to maximal plasma concentration (Tmax)
Pharmacokinetic profile of PRT1419 monotherapy and in combination with AZA or VEN: Area under the curve | Baseline through approximately 3.5 years
  PRT1419 pharmacokinetics will be calculated by area under the plasma concentration x time curve (AUC) from h 0 to the last measurable time point (AUC0-last)
Safety and tolerability of PRT1419 in combination with AZA and VEN: AEs, SAEs, CTCAE assessments | Baseline through approximately 3 years
  Safety and tolerability will be assessed by recording adverse events (AEs), serious adverse events (SAEs), and DLTs according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Anti-tumor activity of PRT1419 monotherapy and in combination with AZA and VEN: Overall response rate (ORR) | Baseline through approximately 3.5 years
  Anti-tumor activity of PRT1419 based on the measurement of objective response rate (ORR) according to the disease-specific response criteria for malignancies under study
Anti-tumor activity of PRT1419 monotherapy and in combination with AZA and VEN: Progression-free survival (PFS)/event free survival (EFS) | Baseline through approximately 3.5 years
  Duration from Day 1 to the earliest date of first disease progression, as assessed by the investigator according to the disease-specific response criteria for malignancies under study, or death due to any cause
Anti-tumor activity of PRT1419 monotherapy and in combination with AZA and VEN: Duration of response (DOR) | Baseline through approximately 3.5 years
  Duration from time of first observed response (CR or PR) to the earliest date of disease progression, as assessed by the investigator according to the disease-specific response criteria for malignancies under study, or death due to any cause
Anti-tumor activity of PRT1419 monotherapy and in combination with AZA and VEN: Overall survival (OS) | Baseline through approximately 3.5 years
  Duration from Day 1 until death due to any cause

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - AdventHealth Bone and Marrow Transplant Center, Orlando, Florida
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - New Jersey Center for Cancer Research, Brick, New Jersey
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - North Shore Hematology Oncology Associates. DBA New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas